CLINICAL TRIAL: NCT01842321
Title: A Phase II Trial Evaluating the Activity of Abiraterone Acetate Plus Prednisone in Patients With a Molecular Apocrine HER2-negative Locally Advanced or Metastatic Breast Cancer
Brief Title: Abiraterone Acetate in Molecular Apocrine Breast Cancer
Acronym: AMA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CADUSEIME02; 2012-002525-29 (EudraCT Number); UC-0140/1206 (Other: UNICANCER)
Record Dates: First submitted 2013-04-24; First posted 2013-04-29 (Estimated); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Breast Cancer
Keywords: locally advanced; metastatic; Breast Cancer; Molecular Apocrine; HER2-negative; Abiraterone acetate
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Abiraterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Abiraterone Acetate (Experimental)
  Interventions: Drug: Abiraterone Acetate

INTERVENTIONS:
Drug: Abiraterone Acetate — Patients will receive abiraterone acetate at 1,000 mg (four 250 mg tablets daily in the morning after an overnight fast) concurrently with prednisone(1) at 10 mg once daily.
  Other Names: ZYTIGA

SUMMARY:
The purpose of this study is to estimate antitumour activity of abiraterone acetate in Patients with a Molecular Apocrine HER2-negative locally advanced or metastatic Breast Cancer.

DETAILED DESCRIPTION:
Screening : All women 18+, with a confirmed locally advanced or metastatic Triple Negative Breast Cancer (TNBC), will be screened and invited to participate (300-500 patients).

Only patients with a centralized confirmation of ER-/PR-/HER2- and evaluation of AR+ will be included and treated with abiraterone acetate plus prednisone (31 patients).

The Treatment phase comprises a series of 4 weeks-cycles with continuous study treatment. Study drug treatment will continue until the earliest of the following events: disease progression, unacceptable toxicity, or death.

At disease progression, patients must be discontinued from study drug and should be evaluated within 30 days during the Post treatment visit and then entered into the Follow-Up phase.Patients should enter the Follow-Up Period regardless of reason for study drug discontinuation and should be monitored every 3 months (± 7 days) during 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Women aged ≥18 years;
* Histologically confirmed locally advanced or metastatic breast cancer;
* Triple negative breast cancer:

Estrogen receptor (ER)-negative and Progesterone receptor (PR)-negative, as defined by a <10 % tumour stained cells by immunohistochemistry (IHC); HER2 negative status (i.e. IHC score 0 or 1+, or IHC score 2+ and FISH/SISH/CISH negative), confirmed centrally before inclusion with FFPE tissue from either primary or metastatic breast cancer site*;

* Androgen receptor (AR)-positive, as defined centrally by a ≥10% tumour stained cells by IHC (AR assessment by local pathologist before inclusion is not mandatory);
* Patients could be chemotherapy naïve (provided they are not presenting with life-threatening metastasis) or have received any number of previous lines of chemotherapy (providing their life expectancy is ≥3 months);
* Pre and post menopausal patients are eligible.
* Measurable or non measurable disease according to RECIST v1.1 criteria;
* PS (ECOG) ≤2;
* Normal haematological function: ANC ≥1,500/mm3; platelets count ≥100,000/mm3; haemoglobin >10 g/dl;
* Normal hepatic function: total bilirubin ≤1.5 upper normal limit (UNL); ASAT and ALAT ≤2.5 UNL (≤5 UNL in the presence of liver metastases);
* Creatinine clearance (MDRD formula) ≥50 mL/min OR creatinine ≤1.5 times ULN;
* Normal kalemia (serum potassium ≥3.5 mM), natremia and magnesemia;
* Systolic blood pressure (BP) <160 mm Hg and diastolic BP <95 mm Hg, as documented on inclusion day (Hypertension at baseline assessment allowed provided it is currently controlled under anti-hypertensive drugs);
* Cardiac ejection fraction ≥50% measured by MUGA or ECHO done within 4 weeks before inclusion;
* If receiving a bisphosphonate or denosumab, dose must have been stable for at least 2 doses before inclusion;
* Patient agreeing to use effective contraception during and for ≥ 6 months after completion of study treatment;
* Patient able to comply with the protocol;
* Patient must have signed a written informed consent form prior to any study specific procedures;
* Patient must be affiliated to a Social Health Insurance.

Exclusion Criteria:

* Male breast cancer;
* HER2-positive status (positivity defined as IHC3+ and/or FISH amplification >2.2);
* Other concurrent malignancies, except adequately treated cone-biopsied in situ carcinoma of the cervix or basal cell or squamous cell carcinoma of the skin; patients who have undergone potentially curative therapy for a prior malignancy are eligible provided there is no evidence of disease for ≥ 5 years and patient is deemed to be at low risk for recurrence;
* Active brain metastases or leptomeningeal disease; History of brain metastases allowed provided lesions are stable for at least 3 months as documented by head CT scan or MRI of the brain;
* Non-malignant systemic disease, including active infection or concurrent serious illness that would make the patient a high medical risk;
* Significant cardiovascular disease, including any of the following:

  1. NYHA class III-IV congestive heart failure;
  2. Unstable angina pectoris or myocardial infarction within the past 6 months;
  3. Severe valvular heart disease;
  4. Ventricular arrhythmia requiring treatment.
* Patients with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption should not be included;
* Patients with known allergies, hypersensitivity or intolerance to abiraterone acetate, prednisone, or their excipients;
* Persistent toxicities ≥ grade 2 from any cause, except chemotherapy-induced alopecia and Grade 2 peripheral neuropathy;
* Active or uncontrolled autoimmune disease requiring concurrent corticosteroid therapy;
* Any gastrointestinal disorder interfering with absorption of the study drug;
* Difficulties with swallowing study capsules;
* Prior anticancer therapy, including radiotherapy, endocrine therapy, immunotherapy, chemotherapy (CT) within the last 3 weeks (2 weeks for oral or weekly CT ; 6 weeks for nitrosoureas and mitomycin C), or other investigational agents ; Concurrent palliative radiotherapy allowed;
* Concurrent enrolment in another clinical trial in which investigational therapies are administered;
* Pregnant women, women who are likely to become pregnant or are breast-feeding;
* Patients with any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial;
* Patients with history of non compliance to medical regimens or unwilling or unable to comply with the protocol;
* Individual deprived of liberty or placed under the authority of a tutor.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2015-07-15 (Actual); Study Completion 2018-07-04 (Actual)

PRIMARY OUTCOMES:
Clinical benefit rate (CBR) | at 6 months
  The 6-months CBR is the measurement of all patients who have a complete response (CR), partial response (PR) or stable disease (SD), according to RECIST criteria v1.1. At six months, patients will be classified as success (Alive at 6 months AND CR/PR/ SD) or failure (dead OR alive with progression).

SECONDARY OUTCOMES:
Objective response rate (ORR) | at 6 months
  The Objective response is defined as complete response (CR) or partial response (PR) according to RECIST criteria v1.1
Duration of overall response (DoR) | at 6 months
  The DoR is defined as the time from documentation of tumour response (CR/PR whichever is first recorded) to disease progression, according to RECIST criteria v1.1.
Overall Survival (OS) | median follow-up = 2 years
  The OS is defined as the time from the first administration of abiraterone acetate to death from any cause.
Progression-free survival (PFS) | median follow-up = 2 years
  The PFS is defined as the time from the first administration of abiraterone acetate to progression or death of any cause, whichever occurs first.
Overall safety profile | during the on-treatment period (defined as the period from the time of first dose of study medications up to 30 days of the last dose)
  The overall safety profile of the treatment is determined by the occurrence of adverse events and toxicities. The severity of the adverse events and toxicities will be graded according the NCI CTCAE scale version 4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Hervé BONNEFOI, Prof., Principal Investigator — Institut Bergonié Bordeaux
Locations (36):
- France (36):
  - Ico - Site Paul Papin, Angers
  - Institut Sainte Catherine, Avignon
  - Chu - Hopital Jean Minjoz, Besançon
  - Institut Bergonie, Bordeaux
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Chu de Brest - Hôpital Morvan, Brest
  - Centre Francois Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Ch Alpes Leman, Contamine-sur-Arve
  - Centre Georges-François Leclerc, Dijon
  - Chu de Grenoble - Hopital Michallon, Grenoble
  - Clinique Sainte Marguerite, Hyères
  - Chd de Vendee, La Roche-sur-Yon
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Ch de Mont de Marsan, Mont-de-Marsan
  - Centre Antoine Lacassagne, Nice
  - Chr D Orleans - Hopital La Source, Orléans
  - Hôpital Saint-Louis, Paris
  - Hôpital Tenon, Paris
  - Institut Curie - Hôpital Claudius Regaud, Paris
  - Ch de Perpignan, Perpignan
  - Ch Lyon Sud, Pierre-Bénite
  - CH de la Région d'Annecy, Pringy
  - Institut Jean Godinot, Reims
  - Centre Henri Becquerel, Rouen
  - Institut Curie - Hôpital René Huguenin, Saint-Cloud
  - Ico- Site Rene Gauducheau, Saint-Herblain
  - Centre Paul Strauss, Strasbourg
  - Hopital Civil - Strasbourg, Strasbourg
  - Hopitaux Du Leman, Thonon-les-Bains
  - Institut Claudius Regaud, Toulouse
  - Ch Bretagne Atlantique, Vannes
  - Hôpital Privé Océane, Vannes
  - Gustave Roussy Cancer Campus, Villejuif

REFERENCES:
- [Derived] Bonnefoi H, Grellety T, Tredan O, Saghatchian M, Dalenc F, Mailliez A, L'Haridon T, Cottu P, Abadie-Lacourtoisie S, You B, Mousseau M, Dauba J, Del Piano F, Desmoulins I, Coussy F, Madranges N, Grenier J, Bidard FC, Proudhon C, MacGrogan G, Orsini C, Pulido M, Goncalves A. A phase II trial of abiraterone acetate plus prednisone in patients with triple-negative androgen receptor positive locally advanced or metastatic breast cancer (UCBG 12-1). Ann Oncol. 2016 May;27(5):812-8. doi: 10.1093/annonc/mdw067. Epub 2016 Feb 18. PMID 27052658